CLINICAL TRIAL: NCT03501238
Title: Interaction and Modulation of Salivary Proteins With Repeat Exposure to Polyphenols
Brief Title: Interaction of Salivary Proteins and Polyphenols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Cordelia Running, PhD, Assistant Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 082-002
Record Dates: First submitted 2017-05-24; First posted 2018-04-18 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Diet Habit; Diet Modification; Taste, Altered; Saliva Altered
MeSH Terms: conditions — Feeding Behavior; Dysgeusia | interventions — Gelatin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know the specifics of each beverage they are taking home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- BSG (Experimental): Participant receives bovine milk, then milk substitute, then milk substitute treated with gelatin
  Interventions: Other: Chocolate Milk; Other: Chocolate milk substitute; Other: Chocolate milk substitute with gelatin
- BGS (Experimental): Participant receives bovine milk, then milk substitute with gelatin, then milk substitute
  Interventions: Other: Chocolate Milk; Other: Chocolate milk substitute; Other: Chocolate milk substitute with gelatin
- SBG (Experimental): Participant receives milk substitute, then bovine milk, then milk substitute with gelatin.
  Interventions: Other: Chocolate Milk; Other: Chocolate milk substitute; Other: Chocolate milk substitute with gelatin
- SGB (Experimental): Participant receives milk substitute, then milk substitute with gelatin, then bovine milk
  Interventions: Other: Chocolate Milk; Other: Chocolate milk substitute; Other: Chocolate milk substitute with gelatin
- GSB (Experimental): Participant receives milk substitute with gelatin, then milk substitute, then bovine milk.
  Interventions: Other: Chocolate Milk; Other: Chocolate milk substitute; Other: Chocolate milk substitute with gelatin
- GBS (Experimental): Participant receives milk substitute with gelatin, then bovine milk, then milk substitute.
  Interventions: Other: Chocolate Milk; Other: Chocolate milk substitute; Other: Chocolate milk substitute with gelatin

INTERVENTIONS:
Other: Chocolate Milk — Chocolate bovine milk will be consumed everyday for 1 week. Milks will be store-bought, with added sucrose and added cocoa powder.
Other: Chocolate milk substitute — Chocolate milk substitute will be consumed everyday for 1 week. Milks will be store-bought, with added sucrose and added cocoa powder.
Other: Chocolate milk substitute with gelatin — Chocolate milk substitute with gelatin added will be consumed everyday for 1 week. Milks will be store-bought, with added sucrose and added cocoa powder.

SUMMARY:
Participants will be chosen through an initial sensory test to find high and low-perceivers of astringency. Selected participants will drink a chocolate milk or milk substitute beverage for one week each with washout weeks in between. At the end of each week participants will taste and rate multiple beverages for their astringency and other sensory properties. Participants will provide saliva samples weekly for proteomic analysis and (potentially) analysis of polyphenols. Participants will also be asked to provide a 24 hour dietary recall once per week. Data will be analyzed to determine if there is a relationship between polyphenol exposure, astringency ratings, and salivary protein composition.

ELIGIBILITY:
Inclusion Criteria:

* High or low perceivers of astringency (from initial screening)

Exclusion Criteria:

* Current smokers (within 30 days), dairy/nut/cocoa allergies, piercings in mouth, mid-range perceiver of astringency, issues with taste, smell, swallowing or choking.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Relative salivary proteins in saliva | 1 year
  Measure relative amounts of salivary proteins in participant saliva.

SECONDARY OUTCOMES:
Subject Diets | 8 months
  Collect participant 24 hour dietary recalls to generate data on eating patterns and dietary choices. Analyze correlations with saliva and sensory ratings. Dietary data that will be analyzed include measures such as: fruit and vegetable intake, fat intake (and type of fat). 24 hour recalls will be assess using the ASHA online tool, which collects data on all foods eaten in the last 24 hours.
Chocolate milk flavor ratings | 8 months
  Measure subjects ratings for astringency, bitterness, sweetness, and liking for chocolate milk. A generalized visual analog scale will be used, ranging from 0 ("None" for intensity and "Worst ever" for liking) to 100 ("Strongest ever" for intensity and "Best ever" for liking).
Chocolate milk substitute flavor ratings | 8 months
  Measure subjects ratings for astringency, bitterness, sweetness, and liking for chocolate almond milk. A generalized visual analog scale will be used, ranging from 0 ("None" for intensity and "Worst ever" for liking) to 100 ("Strongest ever" for intensity and "Best ever" for liking).
Chocolate milk substitute with gelatin flavor ratings | 8 months
  Measure subjects ratings for astringency, bitterness, sweetness, and liking for chocolate almond milk with added gelatin. A generalized visual analog scale will be used, ranging from 0 ("None" for intensity and "Worst ever" for liking) to 100 ("Strongest ever" for intensity and "Best ever" for liking).
Polyphenol content in saliva samples | 8 months
  Measure polyphenol content in expectorated subject saliva samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.